CLINICAL TRIAL: NCT02684565
Title: Effects of Branch Chain Amino Acids on Glucose Tolerance in Obese Pre-Diabetic Subjects
Acronym: BCAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB#15-001928
Record Dates: First submitted 2016-02-09; First posted 2016-02-18 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Prediabetic State
Keywords: pre-diabetes; blood glucose regulation; branching chain amino acids; diabetes; lower blood sugar
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BCAA High Protein supplement (Active Comparator): Subjects will be randomly assigned to take high BCAA protein a day for 4 weeks after a 2-week washout will switch to the other arm.
  Interventions: Dietary Supplement: BCAA High Protein supplement
- BCAA Low Protein Supplement (Active Comparator): Subjects will be randomly assigned to take low BCAA protein a day for 4 weeks after a 2-week washout will switch to the other arm.
  Interventions: Dietary Supplement: BCAA Low Protein supplement

INTERVENTIONS:
Dietary Supplement: BCAA High Protein supplement — Subjects will be randomly assigned to take high BCAA or low-BCAA protein a day for 4 weeks, then switch to BCAA or low-BCAA protein for 4 weeks after a 2-week washout.
  Other Names: INNOBIO Instanized high BCAA Powder
  Arms: BCAA High Protein supplement
Dietary Supplement: BCAA Low Protein supplement — Subjects will be randomly assigned to take high BCAA or low-BCAA protein a day for 4 weeks, then switch to BCAA or low-BCAA protein for 4 weeks after a 2-week washout.
  Other Names: SunWarrior Warrior Blend Natural
  Arms: BCAA Low Protein Supplement

SUMMARY:
Branching chain amino acids (BCAA) have both beneficial and detrimental effects of on metabolism have been established and therefore warrants further investigation. In the preliminary study, the investigators found that BCAAs enhanced glucose metabolism in lean mice while they promoted glucose intolerance in obese mice. In lean mice, BCAAs decreased adiposity and enhanced glucose utilization and insulin sensitivity in different tissues. But in obese mice, BCAAs' effects were mediated by impaired insulin signaling in fat tissue.

This study will examine 10 obese subjects with pre-diabetes and examine the effects of taking BCAA supplement and will monitor the subjects blood glucose, insulin, triglyceride levels and will have an oral glucose tolerance test on repeated occasions to see if any changes are noted in their glucose regulation.

DETAILED DESCRIPTION:
Branched-Chain Amino Acids (BCAAs, including leucine, isoleucine, and valine) regulate multiple cellular functions as nutrient signaling. For example, BCAAs regulate insulin and glucagon secretion and thus glucose metabolism1. BCAAs, especially leucine, is one key regulator of mTOR signaling, which is the central component of a complex signaling network of insulin signaling, cell growth, and proliferation. BCAAs also regulate protein synthesis and degradation in various tissues.

Increasing dietary uptake of BCAAs improved the parameters associated with obesity and T2DM, such as body composition and glycemia levels. However, these beneficial effects are not conclusive. Moreover, other studies have shown that circulating branched-chain amino acid concentrations are associated with obesity and future insulin resistance in children and adolescents.

This is a 12-week, randomized, crossover study with 10 obese subjects with prediabetes. Subjects will be randomly assigned to take 20g BCAA or low-BCAA protein a day for 4 weeks, then switch to BCAA or low-BCAA protein for 4 weeks after a 2-week washout.

At baseline and weeks 4, 6 and 10 weeks glucose, insulin and triglyceride levels will be tested at time 0, 30 min, 60 min, and 120 min after 75 grams of glucose load. In addition to laboratory tests vital signs, weight and body composition will be done.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-50 years of age at screen
2. BMI between 27 to 35
3. Fasting glucose level >100, but <126 mg/dL or HgbA1c >5.7% but < 6.4%
4. Waist circumference > 40 cm in men and >35 in women
5. Subjects must read and sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or enrollment. A subject will be excluded for any condition that might compromise the ability to give truly informed consent.

Exclusion Criteria:

1. Any subject with a history of diabetes mellitus on medications, or other serious medical condition, such as chronic hepatic or renal disease, bleeding disorder, congestive heart disease, cancer (except skin basal cell carcinoma ) chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as systolic BP>160mmHg, diastolic BP>95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, or endocrine diseases (except thyroid disease requiring medication) as indicated by medical history or routine physical examination.
2. Any subject with a screening laboratory value outside of the laboratory normal range that is considered clinically significant for study participation by the investigator.
3. Any subject who currently uses tobacco products.
4. Any history of gastrointestinal disease except for appendectomy.
5. Any antibiotic or laxative use during the 2 months before the study.
6. Any subject who is unable or unwilling to comply with the study protocol.
7. Any subject allergic to soy products.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Change in glucose tolerance composition that Are Related to High protein BCAA Treatment | Baseline to 4 weeks
  The major changes in glucose tolerance after taking supplement
Change in glucose tolerance and body composition that Are Related to Low protein BCAA Treatment | Baseline to 4 weeks
  The major changes in glucose tolerance after taking supplement

SECONDARY OUTCOMES:
Change in glucose tolerance and body composition that Are Related to Low protein BCAA treament | baseline to 4 weeks
  Change in body composition after taking supplement
Change in glucose tolerance and body composition that Are Related to High Protein BCAA treament | Baseline to 4 weeks
  Change in body composition after taking supplement

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD,PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lynch CJ, Adams SH. Branched-chain amino acids in metabolic signalling and insulin resistance. Nat Rev Endocrinol. 2014 Dec;10(12):723-36. doi: 10.1038/nrendo.2014.171. Epub 2014 Oct 7. PMID 25287287
- [Background] McCormack SE, Shaham O, McCarthy MA, Deik AA, Wang TJ, Gerszten RE, Clish CB, Mootha VK, Grinspoon SK, Fleischman A. Circulating branched-chain amino acid concentrations are associated with obesity and future insulin resistance in children and adolescents. Pediatr Obes. 2013 Feb;8(1):52-61. doi: 10.1111/j.2047-6310.2012.00087.x. Epub 2012 Sep 7. PMID 22961720
- [Background] Pal S, Ellis V. The acute effects of four protein meals on insulin, glucose, appetite and energy intake in lean men. Br J Nutr. 2010 Oct;104(8):1241-8. doi: 10.1017/S0007114510001911. Epub 2010 May 11. PMID 20456814